CLINICAL TRIAL: NCT05304169
Title: PRospective, Multicenter Study to Evaluate Safety and Efficacy of Switching Treatments of Prostate Cancer Patients, Initially on Use of Monthly or Quarterly Goserelin Acetate (Zoladex®), to Semiannually Leuprorelin Acetate (Eligard®)
Brief Title: Study to Evaluate the Safety and Efficacy of Switching From Zoladex® Monthly or Quarterly, to Eligard® Semiannual.
Acronym: PRIZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zodiac Produtos Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1500100
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leuprorelin Acetate (Eligard® 45 mg) (Experimental): Patients received two subcutaneous injections of Eligard® 45 mg (leuprorelin acetate), with the first injection given at baseline (Visit 1) and the second after 168 ± 3 days at Visit 4.
  Interventions: Drug: Leuprorelin Acetate (Eligard® 45 mg).

INTERVENTIONS:
Drug: Leuprorelin Acetate (Eligard® 45 mg). — Semiannually Leuprorelin Acetate (Eligard® 45 mg).
  Other Names: Leuprorelin Acetate

SUMMARY:
The purpose of this study is to evaluate the efficacy, quality of life and safety of switching from monthly (3.6 mg) or quarterly (10.8 mg) goserelin acetate (Zoladex®) to semiannual leuprorelin acetate 45 mg (Eligard® 45 mg) in prostate cancer patients with adequate hormonal castration level (plasma testosterone levels ≤50 ng/dL).

DETAILED DESCRIPTION:
When systemic treatment is indicated, androgen deprivation therapy is the standard treatment for patients with prostate cancer. This condition occurs when the patient is diagnosed with metastatic disease or disseminated disease based on PSA values.The exchange of androgen hormone deprivation therapies in patients with metastatic prostate cancer may be required in different situations in clinical practice, such as: lack of medication available at the institution or on the market; alteration of the clinical protocol of the health institution due to economic factors and/or aiming to gain adherence to the treatment, often related to the posological convenience and/or logistics necessary for the administration of the medication, among others.

Additionally, although there is evidence on the efficacy and safety of switching hormone treatments in patients with prostate cancer clinical data on this type of management of patients in Brazil are scarce. There are no data on how the management and switching of treatments is approached, nor on the clinical outcomes related to such a switch of therapy (time to progression, treatments used in combination with androgen deprivation therapy, time to onset of disease symptoms, time to start chemotherapy and costs involved).

ELIGIBILITY:
Inclusion Criteria:

1. Patient able to understand the process of the informed consent form (ICF);
2. Male aged ≥18 years old;
3. Having a histologically confirmed diagnosis of prostate adenocarcinoma;
4. Having an indication of androgen deprivation treatment:

   1. Being on treatment with monthly or quarterly goserelin acetate depot formulation for at least 3 months and for a maximum of 18 months OR;
   2. Having an indication to start treatment with quarterly goserelin acetate depot formulation.
5. Patient with ECOG (Eastern Cooperative Oncology Group) performance status 0 to 2;
6. Patient with appropriate castration level, defined by a serum testosterone level ≤50 ng/dL (≤1.73 nmol/L) demonstrated before V1.
7. Appropriate hematologic function in the screening period: neutrophil count >1,500/μL, platelets >100,000/μL, hemoglobin >10 g/dL;
8. Appropriate liver function in the screening period of the study: total serum bilirubin ≤1.5 x upper normal limit, AST (aspartate aminotransferase) or ALT (alanine aminotransferase) ≤40 U/L, alkaline phosphatase <130 U/L, gamma-GT (glutamyl transferase) <100 U/L;
9. Appropriate kidney function in the screening period of the study: serum urea within normal limits for the method used at the institution, serum creatinine between 0.6 and 1.3 mg/dL, creatinine clearance calculated by the Cockroft- Gault formula > 40 mL/min;

Exclusion Criteria:

1. Patients who did not have or do not have an indication for treatment with goserelin acetate;
2. Patients with goserelin treatment for over 18 months;
3. Patients who have received previous chemotherapy;
4. Patient unable to follow the foreseen study visit schedule;
5. Suspected or proven brain metastasis or active leptomeningeal disease;
6. Uncontrolled arterial hypertension defined as systolic pressure ≥160 mmHg or diastolic pressure ≥95 mmHg;
7. Long-term use of estrogen therapy or peripheral blockade;
8. Another concomitant neoplasm;
9. Any medical condition which, at the investigator's discretion, offers risk to the patient's participation in the study;
10. Having participated in another clinical study within less than 12 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Baseline testosterone levels (≤50 ng/dL) | One year of treatment
  Maintenance of baseline testosterone levels (≤50 ng/dL) after switching from goserelin acetate to leuprorelin acetate 45 mg (Eligard® 45 mg, Zodiac).

SECONDARY OUTCOMES:
Efficacy (consecutive PSA > 4 ng/mL) | One year of treatment
  Disease progression rate from visit 2, defined as 3 consecutive elevations of PSA levels (with PSA > 4 ng/mL) and/or new clinical evidence of disease.
Adverse events frequency (%) | One year of treatment
  Collection and descriptive analysis of adverse events.
Number of Participants With Abnormal Laboratory Values (Number of participants) | One year of treatment
  Determination of the number of participants with abnormal laboratory values defined at discretion of the principal investigator according to reference values. Evaluation of hematologic, kidney and liver function.
Number of Participants With Abnormal Vital Signs (Number of participants) | One year of treatment
  Determination of the number of participants with abnormal vital signs defined at discretion of the principal investigator, according to reference values. Evaluation of vital signs (e.g. electrocardiogram, blood pressure, pulse)
Number of Participants With Abnormal Parameters for Quality of Life according to EORTC QLQ-C30 (Number of Participants) | One year of treatment
  Determination of the number of participants with abnormal parameters for quality of life at discretion of the principal investigator. Quality of life was evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Number of Participants With Abnormal Parameters for Quality of Life according to EORTC QLQ-PR25 (Number of participants) | One year of treatment
  Determination of the number of participants with abnormal parameters for quality of life at discretion of the principal investigator. Quality of life was evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-PR25)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Ferreira Coelho, Principal Investigator — ICESP - Instituto do Câncer do Estado de São Paulo
Locations (6):
- Brazil (6):
  - CPMEC - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - HCB - Hospital do Câncer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - CIP - Centro Integrado de Pesquisa, São José do Rio Preto, São Paulo
  - ICESP - Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo
  - IAMSPE - Instituto de Assistência Médica ao Servidor Público Estadual de S. Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No